CLINICAL TRIAL: NCT02836444
Title: STratification AND Outcome of Patients With the Acute Respiratory Distress Syndrome - A Second Phase Study
Brief Title: Stratification of the Acute Respiratory Distress Syndrome - A Second Phase Study
Acronym: STANDARDS-2
Status: Completed | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Collaborators: Asociación Científica Pulmón y Ventilación Mecánica (Other); Spanish Research Center for Respiratory Diseases (Other)
Responsible Party: Principal Investigator, Jesus Villar, Director, Multidisciplinary Organ Dysfunction Evaluation Research Network, Dr. Negrin University Hospital
Other Study IDs: ACPVM-2015
Record Dates: First submitted 2016-06-23; First posted 2016-07-19 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Current definitions of the Acute Respiratory Distress Syndrome (ARDS) could be adequate for epidemiological studies but are not adequate for inclusion of patients into therapeutic clinical trials. It is a matter of debate whether the assessment of hypoxemia at ARDS onset is appropriate for stratifying lung severity and risk of death in ARDS patients. The investigators will perform an observational, non-interventional, multicenter, prospective audit in a network of intensive care units in Spain for evaluating the severity and risk of death based on the assessment of respiratory and ventilatory function at 24 hours after ARDS diagnosis under standardized ventilatory conditions. This study is the confirmatory phase of the study NCT02288949.

DETAILED DESCRIPTION:
In 2012, an update of the ARDS definition (The Berlin criteria) was published and an empirical classification was proposed according to three PaO2/FiO2 cut-off values at ARDS onset: severe (≤100 mmHg), moderate (>100 - ≤200 mmHg), and mild (>200 - ≤300 mmHg) on positive end-expiratory pressure (PEEP) ≥5 cmH2O. However, despite that there is sufficient evidence about the interactions between PEEP and FiO2, these cut-off values did not mandate the assessment of hypoxemia under standardized guidelines.

The PaO2/FiO2 can be easily manipulated. Alterations in PEEP and FiO2 can dramatically change the PaO2/FiO2. Despite recent reports on the effects of standardized ventilator settings on PaO2/FiO2, is still a matter of debate whether the assessment of hypoxemia must be performed at 24 hours instead of at ARDS onset, and whether the assessment of hypoxemia under standardized ventilator settings is the most appropriate tool for stratifying lung severity in patients with ARDS.

The investigators will examine whether the values of relevant variables (including age, plateau pressure, driving pressure, compliance, PaO2/FiO2) at 24 after ARDS diagnosis under standardized ventilator settings have an impact on the stratification and prediction of death in ARDS patients. This study is an extension of the study NCT02288949.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the Berlin criteria for moderate and severe ARDS.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with moderate and severe ARDS admitted into participating intensive care units, and requiring endotracheal intubation and mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
variables associated with highest and lowest mortality | at 24 hours
  variables associated with highest and lowest mortality

SECONDARY OUTCOMES:
stratification by risk of death | at 24 hours
  stratification by risk of death

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Villar, MD, PhD, Principal Investigator — Hospital Universitario Dr. Negrin
Locations (16):
- Spain (16):
  - Hospital Universitario Mutua de Terrassa, Terrassa, Barcelona
  - Hospital del Bierzo, Ponferrada, León
  - Hospital Universitario NS de Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital Virgen de La Luz, Cuenca
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario de Arrixaca, Murcia
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital General de Segovia, Segovia
  - Hospital Clinico de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Universitario Río Hortega, Valladolid
  - Hospital Virgen de la Concha, Zamora

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Villar J, Gonzalez-Martin JM, Ambros A, Mosteiro F, Martinez D, Fernandez L, Soler JA, Parra L, Solano R, Soro M, Del Campo R, Gonzalez-Luengo RI, Civantos B, Montiel R, Pita-Garcia L, Vidal A, Anon JM, Ferrando C, Diaz-Dominguez FJ, Mora-Ordonez JM, Fernandez MM, Fernandez C, Fernandez RL, Rodriguez-Suarez P, Steyerberg EW, Kacmarek RM; Spanish Initiative for Epidemiology, Stratification and Therapies of ARDS (SIESTA) Network. Stratification for Identification of Prognostic Categories In the Acute RESpiratory Distress Syndrome (SPIRES) Score. Crit Care Med. 2021 Oct 1;49(10):e920-e930. doi: 10.1097/CCM.0000000000005142. PMID 34259448
- [Derived] Villar J, Ambros A, Mosteiro F, Martinez D, Fernandez L, Ferrando C, Carriedo D, Soler JA, Parrilla D, Hernandez M, Andaluz-Ojeda D, Anon JM, Vidal A, Gonzalez-Higueras E, Martin-Rodriguez C, Diaz-Lamas AM, Blanco J, Belda J, Diaz-Dominguez FJ, Rico-Feijoo J, Martin-Delgado C, Romera MA, Gonzalez-Martin JM, Fernandez RL, Kacmarek RM; Spanish Initiative for Epidemiology, Stratification and Therapies of ARDS (SIESTA) Network. A Prognostic Enrichment Strategy for Selection of Patients With Acute Respiratory Distress Syndrome in Clinical Trials. Crit Care Med. 2019 Mar;47(3):377-385. doi: 10.1097/CCM.0000000000003624. PMID 30624279